CLINICAL TRIAL: NCT06368674
Title: Bridging the Gap: Creating a Continuum of Care Through Active Follow-up by a Case Manager After Discharge - a Controlled Study
Brief Title: Bridging the Gap: Creating a Continuum of Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Sahlgrenska University Hospital (Other); Forte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-00363
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Frailty; Dependence; Integrated Care
Keywords: Person-centred care
MeSH Terms: conditions — Frailty | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Clinical control study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group Case Manager (CM) (Experimental): The intervention group will receive extra follow-up by a CM after discharge.
  Interventions: Other: Intervention group Case Manager (CM)
- Control group (Other): The control group will receive usual follow-up after discharge, i.e. no active follow-up
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention group Case Manager (CM) — The CM will be informed about the discharge plan from the nurse at the geriatric ward, as will the municipality for those with need of home help care. An outline of the intervention has been created with managers from primary care and rehabilitation within primary care and municipality care. Core components in the intervention will be active follow-up of the discharge, rehabilitation and care plans. If there are plans that have not been executed or unmet needs, the CM will take adequate contacts to ensure that actions are made to meet the needs. These contacts can be, e.g. the GP for medical needs, the rehabilitation unit in primary or municipality care for unmet rehabilitation needs, and the home help service for unmet care needs. The CM will have a network of contact persons in hospital, primary and community care, as well as in rehabilitation in primary and community care, in order to facilitate for prompt actions to meet the needs.
  Arms: Intervention group Case Manager (CM)
Other: Control Group — The participants in the control group with a planned follow-up by a primary health care centre within the catchment area of the Sahlgrenska University Hospital that does not have CMs designated for active follow up of discharged frail older people. Thus, the participants in the control group will not actively be followed-up after discharge.
  Arms: Control group

SUMMARY:
Coordination and integration between care settings is essential for the quality of care of frail older patients. An active follow-up by a case manager (CM) after discharge form an acute geriatric hospital ward has the potential to bridge the gap between hospital, primary and municipality care for frail older people. This study evaluates the effects of an active follow-up by a CM in primary care after discharge from a geriatric ward, with the following research questions: Can an active follow-up by CM for frail older people discharged from an acute geriatric ward, compared to those not receiving active follow up, Maintain/increase independence in activities of daily living, self-rated health and life satisfaction? Increase satisfaction with health care? Reduce health care consumption/be cost-effective? How feasible is the intervention and the study design from the perspective of the caregivers and the older person? This is a clinical controlled study with a process evaluation. Inclusion criteria are 75 years or older, frail and admitted to a geriatric ward.

This study is relevant since today's highly specialized acute care is poorly adapted to the comprehensive needs of frail older people, and exposes them to avoidable risks such as loss of functional capacities causing unnecessary care needs and decreased wellbeing. Active follow-up by a CM after discharge may be an important way to integrate the care for frail older people, after receiving in-hospital geriatric care. This can improve the quality of care for this vulnerable group, and direct the right health care actions towards those in most need.

The intervention is a active follow-up after discharge by a CM (nurse) in primary care. CM will secure that discharge and care plans are executed and to address new needs. If there are unmet needs, the CM will ensure that adequate actions are performed to meet the needs. The intervention group consists of participants discharged to a primary health care centre with a CM, who actively follows-up after discharge. The control group consists of participants discharged to a primary health care centre without CM, and thereby no active follow-up after discharge. All participants will be followed-up by the research team during one year, concerning dependence in activities of daily living, self-rated health, health care consumption and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

75 years or older, screened as frail, admitted to an acute geriatric ward working according to CGA at the Sahlgrenska or Mölndal hospital. Both hospitals are part of Sahlgrenska University hospital, with the same catchment area, including Gothenburg with surrounding municipalities. People in the region can seek care at both hospitals. The orthopaedic clinic is situated at Mölndal hospital, resulting in most patients with fractures being admitted to this hospital, irrespective of in which municipality they are living. Cognitive impairment is not an exclusion criterion. For people who cannot give informed consent due to cognitive impairment, next of kin will be asked to assist with the consent.

Exclusion Criteria:

Less that 75 years old, Not residing in a permanent residence.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Dependency in Activities of Daily Living (ADL) | Baseline to 12 months
  The primary outcome, dependence in activities of daily living, is measured using the ADL-staircase assessment. It measures dependence in 9 activities: cleaning, shopping, transportation, cooking, bathing, dressing, going to the toilet, transferring, and feeding.
  Dependence is defined as a state in which another person is involved in the activity by giving personal or directive assistance. The sum of dependence in the nine activities of daily living will be calculated, range 0-9, with a clinical significant change of ≥1 unit between baseline and follow up.

SECONDARY OUTCOMES:
Self-rated health | Baseline to 12 months
  Measured by the question: "In general, you would say your health is", with the response alternatives: excellent, very good, good, fair, and poor. Clinically significant difference is ≥1 step in the response alternatives between baseline and follow up.
Life satisfaction | Baseline to 12 months
  Measured using the Fugl-Meyer-Lisat-11questionnaire, which includes 11 items concerning satisfaction with: life as a whole, work, financial situation, leisure, friends and acquaintance, sexual life, functional capacity, family life, partner relationship, physical health, and psychological health. Response alternatives are: very dissatisfied, dissatisfied, rather dissatisfied, rather satisfied, satisfied, and very satisfied. The sum of items for which the respondent reports being satisfied will be calculated, range 0-11, with a clinically significant change of ≥1 between baseline and follow up.
Satisfaction with quality of care | Baseline to 12 months
  Measured by the participants' agreement with the following statements: "I feel that the care given during the hospital stay meets my needs"; "I am satisfied with the hospital care"; "I feel that the care planning meeting before discharge was valuable"; "I was able to take part in the discussions of my needs in the care planning meeting"; "I feel that the actions planned equal my needs", "I feel that the actions delivered equal my needs"; "I feel that the follow-up after discharge by primary care/rehabilitation/ home help care meet my needs"; and "I feel that it is valuable to have a designated case manager in the primary care". The response alternatives are: agree completely, agree partly, neither agree nor disagree, disagree, and disagree completely. An answer of agree completely or agree partly will be considered as being satisfied.
Health economics | 12 months
  Health and social care consumption for 1 year following study enrolment. Health care consumption will be retrieved from the regional care databases, including in-hospital and outpatient care, visits to primary healthcare (physicians, physiotherapists, occupational therapists, nurses, and assistant nurses), and home visits by primary healthcare professionals. The number of readmissions, number of in-hospital days, time to first readmission, and number of outpatient visits will be calculated and compared between intervention and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gothenburg, Gothenburg, Sweden